CLINICAL TRIAL: NCT04955509
Title: In Vivo Optimization and Clinical Application of a Scar Recognition Software for Chronic Spinal Cord Injury (SCI)
Brief Title: A Scar Recognition Software for Chronic Spinal Cord Injury (SCI)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020400，M2020356
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: random splitting based on random sequences generated by engineers to train and optimize a machine learning model
  Interventions: Other: MRI
- Testing: random splitting based on random sequences generated by engineers to evaluate the performance of the model
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — conventional MRI and diffusion MRI

SUMMARY:
To construct and validate a software to recognize scar for patients with chronic SCI based on multimodal MRI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a kind of serious neurologic damage caused by violence to the spinal cord, resulting in various functions of the body below the injury level, including motor, sensory, sphincter, and reflex dysfunction in varying degrees, usually resulting in permanent and irreversible functional loss or paralysis of patients. The treatment of SCI is an essential problem in the world. In the past decades, experimental research on SCI involves genes, proteins, cells, and tissues, and has made great progress. However, these studies mainly focus on the SCI at the early stage, rather than the later stage. The reason is that in the later stage, scar formed by glial cells and fibroblasts in the injured area is a physical and chemical barrier, which inhibits the regeneration and myelination of nerve axons and results in inhibiting spinal cord repairment. Therefore, before the treatment of chronic SCI, the key problem is to distinguish glial scar tissue from normal tissue and eliminate its influence.

As glial scar inhibits axon regeneration, eliminating glial scar is necessary for the repair of the injured spinal cord. In recent years, a large number of experimental studies have been carried out to destroy the process of glial scar formation after SCI by enzyme digestion and antibody. Though these methods reduced glial scar, residual glial scars were reported in animal experiments. Compared to biochemical methods, surgical resection of glial scar tissue is a relatively simple and effective method to eliminate glial scars. Due to the limited regeneration ability of nerves after SCI, it is important to identify scar tissue accurately before operations to avoid surgical injury to normal tissue, which is also the premise of further research and clinical application of various interventional treatment methods.

Magnetic resonance imaging (MRI) is one of the most commonly used non-invasive imaging techniques to evaluate the degree of injury and therapeutic effect of SCI. Nemours MRI studies on SCI show the impact of SCI on the central nervous system from the structural and functional level and prove the potential application value of MRI in assisting doctors in the diagnosis of SCI. A small number of previous studies have used magnetization transfer imaging, and diffusion tensor imaging to detect glial scar tissue, showing the potential application value of these images in differentiation between glial scar and surrounding normal spinal cord. However, because glial cells, which constitute glial scar, are also important components of normal spinal cord tissue, previous studies only identified glial scar from a single aspect, such as tissue type, macromolecular component, or water molecular diffusion strength. Therefore, their specificities were unsatisfactory. Relative methods were unable to identify glial scar accurately and finally resulted in difficulty in treatment arrangement and evaluation of prognosis, which hinders the development of SCI treatment research.

Combing multimodal MRI, including conventional MRI and diffusion MRI, with supervised machine learning makes accurate glial identification in chronic SCI possible. multimodal MRI can depict the differences between scar tissue and non-scar tissue from the aspects of cell composition, water molecular dispersion, structural complexity, etc. Comparing to MRI with a single model, multimodal MRI provides more specific features. Machine learning, a way to construct robust and accurate models, can mine the quantitative relationship between imaging features and clinical diagnosis results, reveal MRI feature markers of the glial scar, to improve the accuracy of identification. The research work, combined with medicine, imaging, and artificial intelligence technology, is expected to solve the problem of accurate and non-invasive identification of glial scar in chronic SCI, which has potential application value for laboratory research and clinical treatment of chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

* (Prospective part) compliance to MRI scan
* (Prospective part) no MRI contraindication
* (Retrospective part) available conventional MRI data
* clinical diagnosis of SCI (the course of disease≥1 year)

Exclusion Criteria:

* prior head or neck surgery or accompanying diseases with neurologic deficits and/or symptoms including multiple sclerosis, motor neuron disease, or spinal cord tumor
* images with motion artifact

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients came from the Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the fitted model | through study completion, an average of 2 year
  positive predictive value (PPV)
Performance of the fitted model | through study completion, an average of 2 year
  sensitivity (SE)
Performance of the fitted model | through study completion, an average of 2 year
  Dice coefficient score (DSC)

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No